CLINICAL TRIAL: NCT01303640
Title: NOBORI Biolimus-Eluting Versus XIENCE/PROMUS Everolimus-eluting Stent Trial
Acronym: NEXT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Professor, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C494
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biolimus-eluting stent (Active Comparator): Biolimus-eluting stent
  Interventions: Device: Biolimus-eluting stent
- Everolimus-eluting stent (Active Comparator): Everolimus-eluting stent
  Interventions: Device: Everolimus-eluting stent

INTERVENTIONS:
Device: Biolimus-eluting stent — Biolimus-eluting stent
  Arms: Biolimus-eluting stent
Device: Everolimus-eluting stent — Everolimus-eluting stent
  Arms: Everolimus-eluting stent

SUMMARY:
The purpose of this study is to evaluate whether the newly-approved biolimus-eluting stent is not inferior to the everolimus-eluting stent in terms of the rate of target-lesion revascularization at 1-year and death or myocardial infarction at 3-year after stent implantation in the real world clinical practice.

DETAILED DESCRIPTION:
Everolimus-eluting stent is the most widely used coronary drug-eluting stent in Japan. Biolimus-eluting stent is a new coronary drug-eluting stent, which is going to be approved in 2011 by the Japanese Ministry of Health, Labor and Welfare. It has been reported that biolimus-eluting stent had lower rate of target-lesion revascularization and stent thrombosis at 9 months as compared with paclitaxel-eluting stent. However, trial results comparing biolimus-eluting stent with everolimus-eluting stent are largely unknown. The purpose of this study is to evaluate whether the newly-approved biolimus-eluting stent is not inferior to the everolimus-eluting stent in terms of the rate of target-lesion revascularization at 1-year and death or myocardial infarction at 3-year after stent implantation in the real world clinical practice. The design of this study is all-comer design enrolling patients scheduled for percutaneous coronary intervention using drug-eluting stents without any exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for percutaneous coronary intervention using drug-eluting stents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3235 (Actual)
Dates: Start 2011-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
target-lesion revascularization | 1-year
  target-lesion revascularization
death or myocardial infarction at 3-year after stent implantation | 3-year
  death or myocardial infarction at 3-year after stent implantation

SECONDARY OUTCOMES:
all-cause death | 3-year
  death due to any cause
cardiac death | 3-year
  death due to cardiac origins
acute myocardial infarction | 3-year
  acute myocardial infarction
stent thrombosis | 3-year
  stent thrombosis defined by Academic Reseach Consortium definition
stroke | 3-year
  stroke excluding transient ischemic attacks
bleeding complications | 3-year
  bleeding complications defined by GUSTO and TIMI definitions
success rate for stent deployment | 3-year
  success rate for stent deployment
procedure time | 3-year
  procedure time
clinically-driven target-lesion revascularization | 3-year
  clinically-driven target-lesion revascularization
non-target-lesion revascularization | 3-year
  non-target-lesion revascularization
coronary artery bypass grafting | 3-year
  coronary artery bypass grafting
target-vessel revascularization | 3-year
  target-vessel revascularization
any repeat coronary revascularization | 3-year
  any repeat coronary revascularization
composite of cardiac death, acute myocardial infarction in the territory of the target vessel or target-lesion revascularization | 3-year
  composite of cardiac death, acute myocardial infarction in the territory of the target vessel or target-lesion revascularization
composite of all-cause death, acute myocardial infarction or any repeat coronary revascularization | 3-year
  composite of all-cause death, acute myocardial infarction or any repeat coronary revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, PhD, Principal Investigator — Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Department of Cardiovascular Medicine, Kyoto University Hospital, Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Ito S, Watanabe H, Morimoto T, Yoshikawa Y, Shiomi H, Shizuta S, Ono K, Yamaji K, Soga Y, Hyodo M, Shirai S, Ando K, Horiuchi H, Kimura T. Impact of Baseline Thrombocytopenia on Bleeding and Mortality After Percutaneous Coronary Intervention. Am J Cardiol. 2018 Jun 1;121(11):1304-1314. doi: 10.1016/j.amjcard.2018.02.010. Epub 2018 Mar 1. PMID 29628128
- [Derived] Watanabe H, Morimoto T, Shiomi H, Yoshikawa Y, Kato T, Saito N, Shizuta S, Ono K, Yamaji K, Ando K, Kaji S, Furukawa Y, Akao M, Ishikawa T, Tamura T, Yamamoto Y, Muramatsu T, Suwa S, Nakagawa Y, Kadota K, Takatsu Y, Nishikawa H, Hiasa Y, Hayashi Y, Miyazaki S, Kimura T. Mortality impact of post-discharge myocardial infarction size after percutaneous coronary intervention: a patient-level pooled analysis from the 4 large-scale Japanese studies. Cardiovasc Interv Ther. 2019 Jan;34(1):47-58. doi: 10.1007/s12928-018-0517-x. Epub 2018 Mar 5. PMID 29508236
- [Derived] Natsuaki M, Kozuma K, Morimoto T, Kadota K, Muramatsu T, Nakagawa Y, Akasaka T, Igarashi K, Tanabe K, Morino Y, Ishikawa T, Nishikawa H, Awata M, Abe M, Okada H, Takatsu Y, Ogata N, Kimura K, Urasawa K, Tarutani Y, Shiode N, Kimura T. Final 3-Year Outcome of a Randomized Trial Comparing Second-Generation Drug-Eluting Stents Using Either Biodegradable Polymer or Durable Polymer: NOBORI Biolimus-Eluting Versus XIENCE/PROMUS Everolimus-Eluting Stent Trial. Circ Cardiovasc Interv. 2015 Oct;8(10):e002817. doi: 10.1161/CIRCINTERVENTIONS.115.002817. PMID 26446596
- [Derived] Natsuaki M, Kozuma K, Morimoto T, Shiomi H, Kimura T. Two-year outcome of a randomized trial comparing second-generation drug-eluting stents using biodegradable or durable polymer. JAMA. 2014 May;311(20):2125-7. doi: 10.1001/jama.2014.3584. No abstract available. PMID 24687156
- [Derived] Natsuaki M, Kozuma K, Morimoto T, Kadota K, Muramatsu T, Nakagawa Y, Akasaka T, Igarashi K, Tanabe K, Morino Y, Ishikawa T, Nishikawa H, Awata M, Abe M, Okada H, Takatsu Y, Ogata N, Kimura K, Urasawa K, Tarutani Y, Shiode N, Kimura T; NEXT Investigators. Biodegradable polymer biolimus-eluting stent versus durable polymer everolimus-eluting stent: a randomized, controlled, noninferiority trial. J Am Coll Cardiol. 2013 Jul 16;62(3):181-190. doi: 10.1016/j.jacc.2013.04.045. Epub 2013 May 15. PMID 23684673